CLINICAL TRIAL: NCT07256483
Title: Influence of the Menstrual Cycle on the Maximal Strength of the External and Internal Rotators of the Shoulder in High-level Sports Women From Montpellier Hérault Rugby.
Brief Title: Influence of the Menstrual Cycle on the Maximal Strength of the External and Internal Rotators of the Shoulder in High-level Sports Women.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A01018-41
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- follicular phase (Experimental): Measures during the follicular phase from D0 to D5
  Interventions: Other: Measure the strength of the external and internal rotator muscles of both shoulders.
- early luteal phase (Active Comparator): Measures during the ovulatory/early luteal phase (approximately days 13 to 18 of the menstrual cycle)
  Interventions: Other: Measure the strength of the external and internal rotator muscles of both shoulders.

INTERVENTIONS:
Other: Measure the strength of the external and internal rotator muscles of both shoulders. — Measure the strength of the external and internal rotator muscles of both shoulders using a Cybex-type isokinetic dynamometer.

SUMMARY:
The goal of this prospective interventional study is to measure the strength of the external and internal rotator muscles of both shoulders (dominant and non-dominant) of Montpellier Hérault Rugby players at different stages of their menstrual cycle. During the menstrual phase (beginning of the follicular phase from D0 to D5) and during the ovulatory/early luteal phase (approximately D13 to D18 of the menstrual cycle). The study is conducted on volunteers.

The main question it aims to answer is : Is there an effect of the menstrual cycle on the maximum strength of the internal and external rotators of the shoulder in female athletes who play rugby?

ELIGIBILITY:
Inclusion Criteria :

* Montpellier Hérault Rugby player
* Regular menstrual cycle
* Adult who has received informed consent information about the study and signed the non-objection form

Exclusion Criteria :

* Use or intake of contraception
* Presence of a condition associated with the menstrual cycle
* Recent injury or pain in the upper limbs lasting more than two weeks, incompatible with performing a test of maximum voluntary contraction of the shoulder rotators
* Presence of an infectious disease (fever) that could skew temperature readings during menstrual cycle monitoring.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Intra-individual correlation of isokinetic torque peaks | baseline and 15 days
  The intra-individual correlation of isokinetic torque peaks (in Nm) measured at two distinct phases of the menstrual cycle (D0-D5 and D13-D18), for each type of internal and external rotator contraction, and for each arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St jean sud de france, Montpellier, France

IPD SHARING:
Plan to Share IPD: No